CLINICAL TRIAL: NCT06044467
Title: A Phase 1B, Repeated Dose Study, to Evaluate the Safety, PD and PK Profile of CM-101 in NAFLD Patients With Normal Liver Function Tests and Stable NAFLD/NASH Patients With NAFLD Activity Score (NAS) < 3-The SPARK Study
Brief Title: The Study of Multiple Doses of CM-101 in Male and Female NAFLD (Nonalcoholic Fatty Liver Disease) and NAFLD/NASH (Nonalcoholic Steatohepatitis) Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-I-002
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anti-human CCL24 monoclonal antibody (CM-101) - study Part One (Experimental): Anti-human CCL24 monoclonal antibody (CM-101)
  NAFLD subjects that have normal liver functions - (Cohort 1: 2.5 mg/kg intravenously and Cohort 2: 5.0 mg/kg subcutaneously)
  Interventions: Drug: Anti-human CCL24 monoclonal antibody (CM-101) - Part One
- Placebo - Study Part One (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo - Study Part One
- Anti-human CCL24 monoclonal antibody (CM-101) - Study Part Two (Experimental): Anti-human CCL24 monoclonal antibody (CM-101)
  NAFLD/NASH patients with NAS < 3 that are in general good health and have normal liver functions - 2.5 mg/kg intravenous infusion
  Interventions: Drug: Anti-human CCL24 monoclonal antibody (CM-101) - Part Two
- Placebo - Study Part Two (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo - Study Part Two

INTERVENTIONS:
Drug: Anti-human CCL24 monoclonal antibody (CM-101) - Part One — Anti-human CCL24 monoclonal antibody (CM-101) - Part One
  Arms: Anti-human CCL24 monoclonal antibody (CM-101) - study Part One
Drug: Anti-human CCL24 monoclonal antibody (CM-101) - Part Two — Anti-human CCL24 monoclonal antibody (CM-101) - Part Two
  Arms: Anti-human CCL24 monoclonal antibody (CM-101) - Study Part Two
Drug: Placebo - Study Part One — Placebo Comparator
  Arms: Placebo - Study Part One
Drug: Placebo - Study Part Two — Placebo Comparator
  Arms: Placebo - Study Part Two

SUMMARY:
A two-part study for NAFLD subjects with normal liver functions and in general good health to be treated with CM-101 or matching placebo and NAFLD/NASH Activity Score (NAS) < 3 that are in general good health and have normal liver functions to be treated with CM-101.

DETAILED DESCRIPTION:
This study is designed to assess the safety and preliminary pharmacodynamics of repeated administrations of CM-101 in two subject populations. The objective of part one of this study is to demonstrate that repeated treatment with CM-101 will be safe and well tolerated in NAFLD subjects that have normal liver functions and are in general good health. A second expansion part will be carried out that will include patients with NAFLD/NASH Activity Score (NAS) < 3 that are in general good health and have normal liver functions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with US confirmation of NAFLD without evidence of NASH;
2. Patients with normal liver function tests (i.e. ALT, AST and ALP).
3. Patients in general good health expected for the preceding 6 months;
4. Women of childbearing potential must agree to use an approved form of contraception prior to study entry and for the duration of study participation through 60 days after the last dose of the study medication. Confirmation that female patients are not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women;
5. Male patients must agree to use a barrier method of contraception or abstinence for the duration of study participation through 60 days after the last dose of the study medication;
6. Patient must be able to read, understand, and sign the informed consent forms (ICF), communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

1. Patients with medical/surgical history of gastric bypass surgery, orthotopic liver transplant (OLT) or patients that are planned for such interventions;
2. Documented history of chronic liver disease (e.g., autoimmune hepatitis (>1:160 ANA with histologic features), Wilson's disease, Hemochromatosis (Ferritin >500 ug/L and percent iron saturation >45%), Primary Biliary Cholangitis, Primary Sclerosing Cholangitis, Alcoholic Liver Disease);
3. Presence of chronic viral hepatitis:

   * Chronic hepatitis B virus (HBV) infection (hepatitis B surface antigen (HBsAg) positive);
   * Chronic hepatitis C virus (HCV) infection (HCV Ab and HCV ribonucleic acid (HCV RNA) positive).

   Patients cured of HCV infection less than 5 years prior to the Screening visit are not eligible;
4. History of or current diagnosis of HCC;
5. Known human immunodeficiency virus (HIV) infection (HIV Ab and HIV ribonucleic acid (HIV RNA) positive);
6. Patients with diabetes mellitus type 1;
7. Patients with uncontrolled diabetes mellitus type 2, i.e. HbA1c ≥ 9% (75 mmol/mol) at the time of screening or patients that are treated with insulin;
8. Patients treated with chronic medication including but not limited to anti-retrovirals, tamoxifen, methotrexate, cyclophosphamide, isotretinoin, bile acid binding resins, or pharmacologic doses of oral glucocorticoids (≥10 mg of prednisone per day or equivalent) within the 12 weeks of screening;
9. Patients treated with the below listed medications can be enrolled into the study if these medications are deemed medically necessary, cannot be stopped and the investigator anticipates their dose will remain stable during the study:

   1. Stable doses of anti-diabetic medications (e.g. metformin, sulfonylureas, SGLT2 inhibitors, glitazones (thiazolidinediones), dipeptidyl peptidase-4 inhibitors and glucagon-like peptide-1 analogs) for at least 6 months prior to screening.
   2. Stable doses of ACE inhibitors, angiotensin II receptor antagonists, beta-blockers and thiazide diuretics for at least 6 months prior to screening.
   3. Stable doses of fibrates, statins, niacin, ezetimibe for at least 6 months prior to screening.
   4. Stable doses of vitamin E for at least 6 months prior to screening.
   5. Replacement therapy (e.g., thyroxine, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed as long as the treatment is stable forat least 6 months prior to screening. For further clarification Insulin treatment is not allowed.
10. Patients with the following medical conditions:

    * Cardiovascular conditions:

      1. Unstable angina (clinical definition)
      2. History of myocardial infarction, cardiac catheterization (for any reason) or coronary artery bypass graft within 18 months of screening
      3. Atrial fibrillation
      4. Congestive Heart failure (clinical definition) or hypertrophic cardiomyopathy
      5. Heart valve disorder (i.e., prosthetic valve or known hemodynamically relevant valve disease)
      6. Unstable angina
    * Uncontrolled thyroid disease
    * Portal hypertension
    * CNS disturbance such as history of Stroke (CVA and/or TIA), Parkinson's disease, Alzheimer's disease, or history of seizure disorders.
    * Autoimmune disease that has required systemic treatment in the 2 years preceding study screening (i.e., with the use of disease-modifying agents, corticosteroids or immunosuppressive drugs).
    * Clinically significant renal dysfunction defined as a serum creatinine concentration >1.4 mg/dL (females) or >1.6 mg/dL (males) and/or a blood urea nitrogen (BUN) concentration >45 mg/dL at screening.
    * Patients diagnosed or treated for any malignancy within 5 years of screening, except in situ malignancy, or low-risk prostate, skin (basal or squamous cell cancer or other localized non-melanoma) or cervix cancer after curative therapy.
    * Any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the patient or impair the assessment of study results.
    * Presence of any condition that could, in the opinion of the investigator, compromise the patient's ability to participate in the study, including a history of substance abuse or a psychiatric condition requiring hospitalization or emergency room visit within 2 years of Screening;
11. Patients with the following blood test abnormalities:

    * Abnormal coagulation tests: INR,
    * Total bilirubin (TB) ≥2 ULN,
    * Serum Albumin < 3.4 g/dL,
    * Platelet count <130 × 10^9/L;
12. History of or current significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day in females and more than 30 g/day in males, on average);
13. Patients with history of substance abuse (including alcohol abuse as defined above) in the past or a positive screen for drugs of abuse (opioids and cannabinoids) or alcohol at screening;
14. Female patients who are pregnant or nursing, or male/female patients who are planning a pregnancy during the course of the study;
15. Patients that are unavailable for follow-up assessments or any concern the investigator may have for patient's compliance with the protocol procedures;
16. Patients that are currently participating or have participated in an interventional clinical study within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence and characteristics of adverse events (AEs) occurring following multiple doses | Up to 18 weeks
  Incidence and characteristics of adverse events (AEs) occurring following multiple doses
Evaluation of the development of anti-drug antibodies (ADA) - Study Part 1 | Up to 18 weeks
  Evaluation of the development of anti-drug antibodies (ADA) following repeated administrations of CM-101 -

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Maximum CM-101 plasma concentration (Cmax) - Study Part 1 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Maximum CM-101 plasma concentration (Cmax)
Plasma Pharmacokinetics (PK) parameters of CM-101 - Time to Cmax (tmax) - Study Part 1 | Up to 18 weeks
  Plasma PK parameters of CM-101 following multiple administrations - Time to Cmax (tmax)
Plasma Pharmacokinetics (PK) parameters of CM-101 - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf - Study Part 1 | Up to 18 weeks
  Plasma PK parameters of CM-101 following multiple administrations - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Terminal elimination rate constant (λz) - Study Part 1 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Terminal elimination rate constant (λz)
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Terminal elimination half-life (T½) - Study Part 1 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Terminal elimination half-life (T½)
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Maximum CM-101 plasma concentration (Cmax) - Study Part 2 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Maximum CM-101 plasma concentration (Cmax)
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Time to Cmax (tmax) - Study Part 2 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Time to Cmax (tmax)
Plasma Pharmacokinetics (PK) parameters of CM-101 following multiple administrations - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf - Study Part 2 | Up to 18 weeks
  Plasma PK parameters of CM-101 - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf
Plasma Pharmacokinetics (PK) parameters of CM-101 - Terminal elimination rate constant (λz) - Study Part 2 | Up to 18 weeks
  Plasma PK parameters of CM-101 following multiple administrations - Terminal elimination rate constant (λz)
Plasma Pharmacokinetics (PK) parameters of CM-101 - Terminal elimination half-life (T½) - Study Part 2 | Up to 18 weeks
  Plasma PK parameters of CM-101 following multiple administrations - Terminal elimination half-life (T½)
Evaluation of the development of anti-drug antibodies (ADA) following repeated administrations of CM-101 - Study Part 2 | Up to 18 weeks
  Evaluation of the development of anti-drug antibodies (ADA) of CM-101
Liver function test: ALT (alanine aminotransferase) - Study Part 2 Only | Over a treatment period of 18 weeks
  Percentage and absolute change from baseline in liver enzymes (liver function test) in multiple timepoints - ALT (alanine aminotransferase)
Liver function test: AST (Aspartate Aminotransferase) - Study Part 2 Only | Over a treatment period of 18 weeks
  Percentage and absolute change from baseline in liver enzymes (liver function test) in multiple timepoints - Liver function test: AST (Aspartate Aminotransferase)
Liver function test: GGT (gamma-glutamyltransferase) - Study Part 2 Only | Over a treatment period of 18 weeks
  Percentage and absolute change from baseline in liver enzymes (liver function test) in multiple timepoints - Liver function test: GGT (gamma-glutamyltransferase)
Liver function test: ALP (Alkaline Phosphatase) - Study Part 2 Only | Over a treatment period of 18 weeks
  Percentage and absolute change from baseline in liver enzymes (liver function test) in multiple timepoints - Liver function test:ALP (Alkaline Phosphatase)
Change from baseline to end of treatment in: fibrosis-4 (FIB-4) score - Study Part 2 Only | Up to 15 Weeks
  Change from baseline to end of treatment in: fibrosis-4 (FIB-4) score
Change from baseline to end of treatment in: Aspartate transaminase (AST) ratio - Study Part 2 Only | Up to 15 Weeks
  Change from baseline to end of treatment in: AST ratio
Change from baseline to end of treatment in: Alanine aminotransferase (ALT) ratio - Study Part 2 Only | Up to 15 Weeks
  Change from baseline to end of treatment in: ALT ratio
Change from baseline to end of treatment in: APRI (AST to platelet ratio index) - Study Part 2 Only | Up to 15 Weeks
  Change from baseline to end of treatment in: APRI (AST to platelet ratio index)
Change from baseline to end of treatment in: Nonalcoholic fatty liver disease (NAFLD) Fibrosis Score - Study Part 2 Only | Up to 15 Weeks
  Change from baseline to end of treatment in: NAFLD Fibrosis Score

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD, Study Chair — ChemomAb Ltd.; Rifaat Safadi, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital - Ein Kerem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mor A, Friedman S, Hashmueli S, Peled A, Pinzani M, Frankel M, Safadi R. Targeting CCL24 in Inflammatory and Fibrotic Diseases: Rationale and Results from Three CM-101 Phase 1 Studies. Drug Saf. 2024 Sep;47(9):869-881. doi: 10.1007/s40264-024-01436-2. Epub 2024 Jun 1. PMID 38822943